CLINICAL TRIAL: NCT00567411
Title: Comparison of the Alpha-2 Agonists for Prevention of Intraocular Pressure Elevation After Selective Laser Trabeculoplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Responsible Party: Vladimir S Yakopson, MD, Ophthalmology Service, Department of Surgery, Walter Reed Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WRAMC WU # 06-23016
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-11

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Laser; laser trabeculoplasty; selective laser trabeculoplasty; intraocular pressure
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Active Comparator): Eyes receiving Apraclonidine 0.5% (Iopidine) prior to SLT
  Interventions: Drug: Apraclonidine 0.5%
- A (Active Comparator): Eyes receiving Brimonidine 0.1% (Alphagan) prior to SLT
  Interventions: Drug: brimonidine 0.1%

INTERVENTIONS:
Drug: brimonidine 0.1% — 1 drop, 1 hour prior to selective laser trabeculoplasty (SLT)
  Arms: A
Drug: Apraclonidine 0.5% — 1 drop applied 1 hour prior to SLT
  Arms: I

SUMMARY:
The purpose of the study is to compare the safety and efficacy of two drops used to lower eye pressure when given prior to a glaucoma laser procedure.

DETAILED DESCRIPTION:
This is a prospective randomized double blind trial of patients undergoing selective laser trabeculoplasty for primary open angle glaucoma and ocular hypertension. Enrolled patients are randomized to receive one drop of brimonidine 0.1% in one eye and one drop of apraclonidine 0.5% in the fellow eye. The trabecular meshwork in both eyes of each enrolled patient is treated 360 degrees at the same sitting. Intraocular pressure is measured in each eye one hour before applying the study medications and at one hour and one week after laser surgery.

ELIGIBILITY:
Inclusion Criteria:

* male or female, at least 18 years of age
* Open Angle Glaucoma with inadequate intraocular pressure (IOP) control or evidence of progression (based on optic nerve head appearance and/or visual field changes) despite current medical therapy
* Ocular Hypertension requiring lowering of IOP
* ability to understand and provide informed consent to participate in this study and willingness to follow study instructions and likely to complete all required visits

Exclusion Criteria:

* inability to understand and provide informed consent to participate in this study
* inability/unwillingness to follow study instructions and complete all required visits
* Documented allergy to either brimonidine or iopidine
* Angle Closure Glaucoma
* Congenital/Juvenile Glaucoma
* Neovascular Glaucoma
* Active uveitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2006-08; Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative IOP | 1 hour and 1 week post surgery

SECONDARY OUTCOMES:
Overall IOP reduction post SLT | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir S Yakopson, MD, Principal Investigator — Walter Reed AMC
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States